CLINICAL TRIAL: NCT05840549
Title: A Randomised Feasibility Study COmparing Urolift and Standard Transurethral Resection of Prostate Ahead of Radiotherapy in Men With Urinary Symptoms Secondary to Prostate Enlargement
Brief Title: A Study Comparing Urolift and TURP Ahead of Radiotherapy in Men With Urinary Symptoms Secondary to Prostate Enlargement
Acronym: CO-STAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: King's College London (Other); St George's University Hospitals NHS Foundation Trust (Other); Institute of Cancer Research, United Kingdom (Other); North Cumbria University Hospitals NHS Trust (Other); University College, London (Other); City, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CCR5668
Record Dates: First submitted 2023-01-17; First posted 2023-05-03 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TURP (Active Comparator): Transurethral Resection of Prostate
  Interventions: Procedure: TURP
- UroLift (Experimental): UroLift
  Interventions: Procedure: UroLift

INTERVENTIONS:
Procedure: TURP — TURP is an operation which can be performed under a general / regional anaesthetic. A cystoscope is passed into the urethra meatus, along the length of the urethra to the level of the prostate. The obstructing prostate lobes are resected using mono polar or bipolar energy to create a channel for improved urinary flow. Haemostasis is achieved by coagulation followed by insertion of a catheter for irrigation post procedure. Generally, patients stay for 1-2 nights post operatively. On the day of discharge the catheter is removed.
  Arms: TURP
Procedure: UroLift — UroLift (Neotract) is a NICE-approved alternative to TURP that can be performed under local anaesthetic, sedation or general anaesthetic. The system comprises of two single-use components, a delivery device and an implant. The implant is made of a nitinol capsular tab, a polyethylene terephthalate monofilament and a stainless-steel end-piece. Again, a modified cystoscope is passed into the urethral meatus, along the length of the urethra to the level of the prostate. The delivery device deploys the implants into the prostate to 'pin' back the lobes of the prostate to create a channel for improved flow. Typically, 2-4 implants are used per procedure. Nine out of ten patients do not require a catheter post procedure
  Arms: UroLift

SUMMARY:
Prostate cancer affects 1 in 8 men and in the UK approximately 14,000 men are treated with radiotherapy.

Around half of men diagnosed with prostate cancer will also have an enlarged prostate making it difficult to pass urine. When having radiotherapy, the prostate swells further which can lead to complete blockage of urine flow (urine retention), sepsis and kidney failure in severe cases. Radiotherapy itself can also cause urinary symptoms meaning that some patients can continue to have difficulty passing urine long after their cancer treatment finishes. Around a third of patients will need an operation to shrink their prostate before radiotherapy to prevent these possible short and long-term problems.

The standard operation is a transurethral resection of prostate (TURP). This involves cutting a channel through the prostate to improve urine flow.

This will be compared with a newer procedure known as UroLift. During UroLift, clips are inserted into the water pipe to pin back the prostate to widen the channel and improve urine flow. Which treatment is more acceptable to patients and gives better outcomes has never been tested before in men having radiotherapy for prostate cancer.

The study will help us to understand how the treatments impact on a patient's quality of life and understand what matters most to patients.

The results of this feasibility study will help us design a bigger study to assess TURP and UroLift in a larger group of patients across different hospitals. This research will help future patients make decisions about prostate cancer treatment choices that can affect their long-term well-being.

DETAILED DESCRIPTION:
Prostate radiotherapy can cause lower urinary tract symptoms (LUTS) such as urinary frequency, difficulty starting a urine stream or feelings of incomplete emptying. 50% of men aged over 60 years may have pre-existing LUTS from bladder outflow obstruction (BOO) due to prostatic enlargement.

The short-term complications of untreated BOO in the context of prostate radiotherapy, although relatively rare, can be disastrous, leading to urinary retention, sepsis and renal failure. In the long-term, urinary symptoms and complications can continue to worsen. Patients with low flow rates pre-radiotherapy are at highest risk of urinary retention and are often offered transurethral resection of prostate (TURP) prior to radiotherapy. An urgent transurethral resection of prostate (TURP) either during or post radiotherapy may significantly disrupt the completion of the treatment and compromise outcomes, both oncological and functional. Case studies suggest that when patients undergo a TURP to treat prostate enlargement after radiotherapy, the risk of incontinence is much higher than surgery before radiotherapy. Therefore, for radiotherapy to safely go ahead, BOO due to an enlarged prostate must first be addressed. UroLift is a newer, minimally invasive alternative to TURP, approved by NICE for use in BPH and available in over 100 trusts nationally. A growing body of evidence including three meta-analyses supports its use in benign disease.

UroLift has not been trialled in patients undergoing prostate radiotherapy with coexisting LUTS. A subgroup analysis performed on retrospective data suggested that patients who had previously undergone prostate radiotherapy experienced symptom relief without an increase in adverse events.

The purpose of this trial is to produce a protocol for a randomised controlled evaluation of clinical and cost effectiveness of UroLift in comparison to TURP for men due to receive radiotherapy as treatment for prostate cancer. At the end of this study, we will understand whether such a trial is acceptable to all stakeholders, is methodologically robust and thus feasible. Furthermore, we will be able to report pilot findings for safety and efficacy

ELIGIBILITY:
Inclusion Criteria:

* Men undergoing prostate radiotherapy for prostate cancer
* Patients with moderate to severe and/or bothersome lower urinary tract symptoms secondary to prostate enlargement and/or an obstructive flow rate
* Patients willing and able to provide written informed consent for the study.

Exclusion Criteria:

* Extensive locally advanced disease
* Unfavourable anatomical features (e.g. large middle lobe, for UroLift this requires advanced techniques that have not been fully evaluated in the benign setting(11)
* Prostates over 100g (as per manufacturer's guidelines)
* Co-morbidities precluding surgical intervention
* Prior prostate cancer treatment (including radical prostatectomy, focal therapy i.e. brachytherapy / high intensity focal ultrasound)
* Prior surgical intervention for benign prostatic hyperplasia (including prior UroLift / TURP / other prostate de-obstructing procedures)
* Urinary symptoms not due to prostatic enlargement as primary cause (i.e. neurological disease)
* Patients with complications of prostate enlargement including catheter dependent retention, recurrent urinary tract infections, bladder stones, obstructive uropathy
* Urinary incontinence due to an incompetent sphincter
* Co-existing gross haematuria
* Current active urinary tract infection

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-05-09 (Estimated); Study Completion 2025-05-09 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate (number of patients enrolled) | Number of patients recruited measured at 3 months
  We will evaluate whether it is possible to recruit patients to an RCT comparing standard treatment with a new treatment untested in the cancer arena
Recruitment rate (number of patients enrolled) | Number of patients recruited measured at 6 months
  We will evaluate whether it is possible to recruit patients to an RCT comparing standard treatment with a new treatment untested in the cancer arena
Recruitment rate (number of patients enrolled) | Number of patients recruited measured at 9 months
  We will evaluate whether it is possible to recruit patients to an RCT comparing standard treatment with a new treatment untested in the cancer arena
Recruitment rate (number of patients enrolled) | Number of patients recruited measured at 12 months
  We will evaluate whether it is possible to recruit patients to an RCT comparing standard treatment with a new treatment untested in the cancer arena
Retention rate | End of study (24 months)
  We will assess the proportion of patients who will complete the trial protocol

SECONDARY OUTCOMES:
Acceptability of intervention | End of study (24 months)
  The Research Team will carry out 12 in-depth interviews. Using the Theoretical Framework of Acceptability(19), affective attitudes, burden, ethicality, intervention coherence, opportunity costs and perceived effectiveness will be assessed
Change from baseline in patient reported outcomes as assessed by the Extended Prostate Cancer Index Composite-50 (EPIC-50) | Baseline, 6 weeks and three months post intervention
  The EPIC-50 is a validated questionnaire for measuring health related quality of life
Change from baseline in patient reported outcomes as assessed by the UCLA Prostate Cancer Index (UCLA-PCI) | Baseline, 6 weeks and three months post intervention
  The UCLA-PCI is a validated questionnaire for measuring health related quality of life
Change from baseline in patient reported outcomes as assessed by the International Consultation on Incontinence Questionnaire-Urinary Incontinence (ICIQ-UI) | Baseline, 6 weeks and three months post intervention
  The ICIQ-UI is a validated questionnaire s a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence
Change from baseline in patient reported outcomes as assessed by the EuroQol EQ-5D | Baseline, 6 weeks and three months post intervention
  The EQ-5D is a validated questionnaire for measuring health related quality of life
Change from baseline in patient reported outcomes as assessed by the Couples Illness Communication Scale (CICS) | Baseline, 6 weeks and three months post intervention
  The CICS is a validated questionnaire for assessing illness-related couple communication
Change post surgery & post radiotherapy in patient reported outcomes as assessed by the patient global impression of improvement (PGI) | 6 weeks and three months post intervention
  The PGI is a validated single item self reported scale to assess patient reported post-operative improvement in condition
Change from baseline in patient reported outcomes as assessed by the International Prostate Symptom Score (IPSS) | Baseline, 6 weeks and three months post intervention
  The IPSS is a validated questionnaire for measuring the severity of urinary symptoms and overall quality of life
Post treatment functional assessment of cancer therapy prostate (FACT-P) | Three months post intervention
  The FACT-P is a multidimensional, self-reported quality of life instrument consisting of 27 core items that assess participant function in 4 domains: physical, social/family, emotional, functional well-being, and supplemented by 12 site-specific items to assess for prostate-related symptoms. Each item is rated on a 0 to 4 Likert-type scale, and then combined to produce subscale scores for each domain. Total subscale score range for physical well-being domain is from 0 (worst response) to 28 (best response), where higher score indicate better quality of life.
Health related quality of life questionnaires | End of study (24 months)
  collected and assessed for appropriateness, usability and completeness for both arms 3 months post radiotherapy treatment
Safety | 30 days post surgery
  30 day surgical morbidity rates will be collected with respect but not limited to infection, urinary retention and bleeding.
Efficacy of procedure | End of study (24 months)
  Improvement in baseline IPSS score
Efficacy of procedure | End of study (24 months)
  Improvement in baseline Urine flowmetry (measured by increased maximum flow rate)
Efficacy of procedure | End of study (24 months)
  Improvement in baseline Urine flowmetry (measured by post void residual)
Cost of intervention | End of study (24 months)
  Information on costs of the two interventions
Re-Operation rate | End of study (24 months)
  Rate of re-operation for technical failure to reduce outflow obstruction

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - St Georges University Hospital, London, Lon
  - Kathie Wong, Carlisle
  - The Royal Marsden NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong K, Kinsella N, Seth J, Nicol D, Cahill D, Kasivisvanathan R, Withington J, Moghul M, Moss CL, Van Hemelrijck M, Giorgakoudi K, Cottrell C, Yates E, Khoo V, James ND. COmparing Urolift and Standard Transurethral resection of prostate Ahead of Radiotherapy in men with urinary symptoms secondary to prostate enlargement in Southwest London and North Cumbria (CO-STAR): a study protocol for a randomised feasibility study. BMJ Open. 2023 Oct 6;13(10):e076621. doi: 10.1136/bmjopen-2023-076621. PMID 37802612